CLINICAL TRIAL: NCT03521375
Title: VIdeo Assisted Thoracoscopic Lobectomy Versus Conventional Open LobEcTomy for Lung Cancer, a Multi-centre Randomised Controlled Trial With an Internal Pilot
Brief Title: VIdeo Assisted Thoracoscopic Lobectomy Versus Conventional Open LobEcTomy for Lung Cancer
Acronym: VIOLET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bristol (Other)
Collaborators: Royal Brompton & Harefield NHS Foundation Trust (Other); University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ORCA58877
Record Dates: First submitted 2018-01-26; First posted 2018-05-11 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Lung Neoplasms
Keywords: lung; cancer; lobectomy
MeSH Terms: conditions — Lung Neoplasms; Neoplasms | interventions — Conversion to Open Surgery; Thoracic Surgery, Video-Assisted

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VATS lobectomy (Experimental): VATS lobectomy is undertaken through one to four keyhole incisions without rib spreading. The use of 'rib spreading' is prohibited as this is the key intra-operative manoeuvre which disrupts tissues and causes pain (and is used in open surgery). The procedure is performed with videoscopic visualisation without direct vision. The hilar structures are dissected, stapled and divided. Endoscopic ligation of pulmonary arterial branches may be performed. The fissure is completed and the lobe of lung resected. Lymph node management is the same as described for open surgery. The incisions are closed in layers and may involve muscle, fat and skin layers. This definition of VATS lobectomy is a modification of CALGB 39802.
  Interventions: Procedure: Video Assisted Thoracoscopic Surgery (VATS)
- Open lobectomy (Active Comparator): Conventional open surgery is undertaken through a single incision +/- rib resection and with rib spreading. The operation is performed under direct vision with isolation of the hilar structures (vein, artery and bronchus) which are dissected, ligated and divided in sequence and the lobe of lung resected. The procedures may be undertaken using ligatures, over sewing or with staplers. Lymph node management is undertaken in accordance with the International Association of the Study of Lung Cancer (IASLC) recommendations where a minimal of 6 nodes / stations are removed, of which 3 are from the mediastinum that includes the subcarinal station. The thoracotomy is closed in layers starting from pericostal sutures over the ribs, muscle, fat and skin layers.
  Interventions: Procedure: Open Surgery

INTERVENTIONS:
Procedure: Open Surgery — Conventional open surgery is undertaken through a single incision +/- rib resection and with rib spreading. The operation is performed under direct vision with isolation of the hilar structures (vein, artery and bronchus) which are dissected, ligated and divided in sequence and the lobe of lung resected. The procedures may be undertaken using ligatures, over sewing or with staplers. Lymph node management is undertaken in accordance with the International Association of the Study of Lung Cancer (IASLC) recommendations where a minimal of 6 nodes / stations are removed, of which 3 are from the mediastinum that includes the subcarinal station. The thoracotomy is closed in layers starting from pericostal sutures over the ribs, muscle, fat and skin layers.
  Other Names: Open lobectomy
  Arms: Open lobectomy
Procedure: Video Assisted Thoracoscopic Surgery (VATS) — VATS lobectomy is undertaken through one to four keyhole incisions without rib spreading. The use of 'rib spreading' is prohibited as this is the key intra-operative manoeuvre which disrupts tissues and causes pain (and is used in open surgery). The procedure is performed with videoscopic visualisation without direct vision. The hilar structures are dissected, stapled and divided. Endoscopic ligation of pulmonary arterial branches may be performed. The fissure is completed and the lobe of lung resected. Lymph node management is the same as described for open surgery. The incisions are closed in layers and may involve muscle, fat and skin layers. This definition of VATS lobectomy is a modification of CALGB 39802.
  Other Names: VATS lobectomy
  Arms: VATS lobectomy

SUMMARY:
Lung cancer is the leading cause of cancer death worldwide and survival in the United Kingdom (UK) remains amongst the lowest in Europe. Surgery is the main method of managing early stage disease and is traditionally undertaken via conventional open surgery. However, over the last decade there has been a surge in the number of minimal access resections performed using Video-assisted thoracoscopic surgery (VATS). However, there remains a need for well-designed and conducted randomised controlled trial (RCT) to provide the evidence base for the wide spread uptake and delivery of this surgical approach.

DETAILED DESCRIPTION:
The uptake of surgery for lung cancer in the UK is low and minimal access surgery may be regarded as a more acceptable intervention (compared to open surgery) by patients, referring respiratory physicians and oncologists. However, a large multi-centre RCT is essential to inform patient and clinician decision making and influence surgical practice in the UK.

The VIOLET study will compare the effectiveness, cost-effectiveness and acceptability of VATS lobectomy versus open surgery for treatment of lung cancer and will test the hypothesis that VATS surgery is superior to open surgery with respect to self-reported physical function five weeks after randomisation (approx. one month after surgery).

Specific objectives are to estimate:

A. The difference between groups in the average self-reported physical function at five weeks.

B. The difference between groups with respect to a range of secondary outcomes including assessment of efficacy (hospital stay, pain, proportion and time to uptake of chemotherapy), measures of safety (adverse health events), oncological outcomes (proportion of patients upstaged to pN2 disease and disease free survival) and overall survival.

C. The cost effectiveness of VATs and open surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged ≥16 years of age
2. Able to give written consent, undergoing either:

   i. Lobectomy or bilobectomy for treatment of known or suspected primary lung cancer beyond lobar orifice* in TNM8 stage cT1-3 (by size criteria, equivalent to TNM7 stage cT1a-2b) or cT3 (by virtue of 2 nodules in the same lobe), N0-1 and M0 or ii. Undergoing frozen section biopsy with the intention to proceed with lobectomy or bilobectomy if primary lung cancer with a peripheral tumour beyond a lobar orifice* in TNM8 stage cT1-3 (by size criteria, equivalent to TNM7 stage cT1a-2b) or cT3 (by virtue of 2 nodules in the same lobe), N0-1 and M0 is confirmed
3. Disease suitable for both minimal access (VATS) and open surgery

Exclusion Criteria:

1. Adults lacking capacity to consent
2. Previous malignancy that influences life expectancy
3. Patients in whom a pneumonectomy, segmentectomy or non-anatomic resection (e.g. wedge resection) is planned
4. Patients with a serious concomitant disorder that would compromise patient safety during surgery.
5. Planned robotic surgery

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 503 (Actual)
Dates: Start 2015-07; Primary Completion 2019-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Self-reported physical function using HRQoL questionnaire QLQ-C30 | 5 weeks post randomisation
  Physical functioning scale, ranges between 0 and 100. High score indicates high level of physical functioning.

SECONDARY OUTCOMES:
Time from surgery to hospital discharge, assessed up to 12 months | Time from surgery to hospital discharge, assessed up to 12 months
Adverse health events to 1 year | Adverse health events to 1 year
Proportion of patients taking up adjuvant treatment, assessed up to 12 months | Proportion and time to uptake of adjuvant treatment, assessed up to 12 months
Time to uptake of adjuvant treatment, assessed up to 12 months | Proportion and time to uptake of adjuvant treatment, assessed up to 12 months
Proportion of patients upstaged to pN2 disease after surgical procedure, assessed up to 3 months post surgery | Proportion of patients upstaged to pN2 disease after surgical procedure, assessed up to 3 months post-surgery
Overall and disease-free survival to 1-year | 1 year
Proportion of patients who undergo complete resection during the procedure, , assessed up to 12 months | Proportion of patients who undergo complete resection during the procedure, assessed up to 12 months
Proportion of patients who experience prolonged incision pain (defined as the need of analgesia > 5 weeks post-randomisation) | Up to 1 year
Disease-specific HRQoL - EORTC QLQ-C30 to 1-year | Measured at 2 week, 5 weeks, 3 months, 6 months and 1-year post randomisation
  3 types of scales. Functioning scales which include physical functioning, role functioning, emotional function, cognitive functioning and social functioning. Symptom scales which include fatigue, nausea and vomiting, pain, dysponea, insomnia, appetite loss, constipation, diarrhoea, financial difficulties.
  An overall global health status/QoL All scales range between 0 and 100. For functioning scales, a high score indicates a high level of functioning. Similarly, a high global health status/QoL score indicates a high quality of life. For symptom scales, a high score indicates a high level of symptoms.
Disease-specific HRQoL - EORTC QLQ-LC13 to 1-year | Measured at 2 week, 5 weeks, 3 months, 6 months and 1-year post randomisation
  Symptoms scales which include Dyspnoea, Couging, Haemoptysis, Sore mouth, Dysphagia, Peripheral neuropathy, Alopecia, Pain in chest, Pain in arm or shoulder, Pain in other parts, and Pain medication. For these scales, a high score indicates a high level of symptoms, as with the QLQ-C30.
  Scales range between 0 and 100.
Generic HRQoL - EORTC EQ5D to 1-year | Measured at 2 week, 5 weeks, 3 months, 6 months and 1-year post randomisation
  Subscales: mobility, self-care, usual activities, pain/discomfort, anxiety/depression. These range from 1-5.
  subscales mobility, self-care, usual activities, pain/discomfort, anxiety/depression are combined to calculate an overall index score which ranges from -0.59 to 1.
  A higher score indicates better quality of life
Resource use | Up to 1 year
  Resource use to 1-year (measured for the duration of post-operative hospital stay until discharge, and at 5 weeks, 3 months, 6 months and 1-year post randomisation)

CONTACTS AND LOCATIONS:
Overall Officials: Chris Rogers, Study Director — University of Bristol; Eric Lim, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust
Locations (9):
- United Kingdom (9):
  - Heartlands Hospital, Birmingham
  - Bristol Royal Infirmary, Bristol
  - Royal Infirmary of Edinburgh, Edinburgh
  - Hull and East Yorkshire Hospitals NHS Trust, Hull
  - Liverpool Heart and Chest Hospital NHS Foundation Trust, Liverpool
  - Harefield Hospital, London
  - Royal Brompton Hospital, London
  - The James Cook University Hospital, Middlesbrough
  - Oxford University Hospitals NHS Foundation Trust, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lim E, Batchelor T, Shackcloth M, Dunning J, McGonigle N, Brush T, Dabner L, Harris R, Mckeon HE, Paramasivan S, Elliott D, Stokes EA, Wordsworth S, Blazeby J, Rogers CA; VIOLET Trialists. Study protocol for VIdeo assisted thoracoscopic lobectomy versus conventional Open LobEcTomy for lung cancer, a UK multicentre randomised controlled trial with an internal pilot (the VIOLET study). BMJ Open. 2019 Oct 14;9(10):e029507. doi: 10.1136/bmjopen-2019-029507. PMID 31615795
- See also: Protocol paper publication — https://bmjopen.bmj.com/content/9/10/e029507.citation-tools